CLINICAL TRIAL: NCT02597335
Title: Non Invasive IDentification of Gliomas With IDH1/2 Mutation by Analysis of Circulating Plasmatic DNA, D-2-hydroxyglutarate Dosage in Biological Liquids and Detection by Brain SPEctro-MRI: Impact for Diagnosis and Follow-up
Brief Title: Non Invasive Detection of IDH1/2 Mutation in Gliomas
Acronym: IDASPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120141
Record Dates: First submitted 2015-04-27; First posted 2015-11-05 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2016-12

CONDITIONS: Glioma; IDH1/IDH2 Mutation
Keywords: Glioma; IDH1/IDH2 mutation; Spectroscopy MRI; D-2-hydroxyglutarate; Free circulating DNA
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IDH1/IDH2 (Experimental)
  Interventions: Radiation: Spectro-MRI; Other: Dosage of free circulating plasmatic DNA; Other: Dosage of D-2HG in the urine

INTERVENTIONS:
Radiation: Spectro-MRI — Spectro-MRI for D-2HG detection
Other: Dosage of free circulating plasmatic DNA
Other: Dosage of D-2HG in the urine

SUMMARY:
This trial develops a non invasive diagnostic approach of IDH1 mutated gliomas combining mutation detection from free plasmatic DNA, D-2HG dosage in urine samples, and D-2HG detection by Brain Spectro MRI.

In group 1 (25 patients), patients with presumed grade II-III gliomas candidate to surgery will undergo spectro MRI, plasma, urine dosages. Results will then be confronted to tumor mutational status and D-2HG.

In group 2 (15 patients), patients with known IDH1 mutation will undergo spectro MRI, plasma, urine dosages overtime in order to correlate results with the response to treatment.

DETAILED DESCRIPTION:
The aim of this trial is to develop and validate a non invasive diagnostic approach of IDH1 mutated gliomas. It will evaluate the specificity and sensitivity of D-2HG detection by Brain Spectro MRI. This approach will be coupled with mutation detection from free plasmatic DNA and D-2HG dosage in urine samples.

The primary end-point is the quantification of D-2HG by spectro-MRI, and the correlation with the dosage of D-2HG in the tumor fragment, and the mutational status (group 1: 25 patients).

The secondary endpoints include:

1. longitudinal analysis Spectro-MRI overtime (12 months) correlation with radiological evolution and the response to treatment (group 2: 15 patients)
2. Differentiation of tumor recurrence from radiation induced changes
3. Confrontation of Spectro-MRI, D-2HG dosages and IDH mutation detection from plasma DNA, and elaboration of a combined score of prediction

ELIGIBILITY:
Inclusion criteria

1. Affiliation to a social security system
2. Patient≥ 18 years old
3. Written informed consent
4. One of the two situations:

   * presumed grade II-III glioma candidate to surgery (group 1)
   * IDH1/IDH2 mutated grade II-III gliomas, candidate to chemotherapy or radiotherapy treatment, or simple follow-up (group 2)
5. Evaluable tumoral mass min diameter >2 cm (FLAIR)
6. PKPS > 60

Exclusion criteria

1. Contra-indication to MRI
2. Patient unable to give an written Informed Consent
3. Patient under guardianship or deprived of freedom
4. For group 2: patient already included in group 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
D-2HG quantified by spectroMRI the measure of the ratio between two pics D-2HG and creatine [Time Frame: 3 months after surgery] [Designated as safety issue: No] | 3 months after surgery
  This ratio D-2HG/creatine will be correlated with the dosage obtained in tumor tissue performed within three months after the surgery

SECONDARY OUTCOMES:
SpectroMRI [Time Frame: evolution over 12 months] [Designated as safety issue: No] | evolution over 12 months
  The ratio D-2HG/creatine will be evaluated overtime and correlated with radiological evolution and the response to treatment (group 2: 15 patients) every four months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sanson, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France